CLINICAL TRIAL: NCT05776914
Title: Efficacy and Safety of Proteolytic Activity-Guided Fecal Microbiota Transplantation for Irritable Bowel Syndrome (PRAGMAT Trial)
Brief Title: Fecal Microbiota Transplantation for IBS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Madhusudan (Madhu) Grover, MBBS (Other)
Responsible Party: Sponsor-Investigator, Madhusudan (Madhu) Grover, MBBS, Regulatory Sponsor and Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-005385
Record Dates: First submitted 2023-03-01; First posted 2023-03-20 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Irritable Bowel Syndrome; Diarrhea
Keywords: Post-infection irritable bowel syndrome with diarrheal; Post-infection irritable bowel syndrome with mixed symptoms
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donor Fecal Microbiota Transplantation Group (Experimental): Subjects will receive a fecal microbiota transplantation (FMT) using stool from a donor
  Interventions: Biological: Donor Fecal Microbiota Transplantation
- Autologous Fecal Microbiota Transplantation Group (Placebo Comparator): Subjects will receive a fecal microbiota transplantation (FMT) using their own stool
  Interventions: Biological: Autologous Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Donor Fecal Microbiota Transplantation — Single fecal microbiota transplantation using 50 gm of freeze-thawed donor stool
  Arms: Donor Fecal Microbiota Transplantation Group
Biological: Autologous Fecal Microbiota Transplantation — Single fecal microbiota transplantation using 50 gm of stool collected from the same individual
  Arms: Autologous Fecal Microbiota Transplantation Group

SUMMARY:
The purpose of this study is to learn the efficacy and safety of fecal microbiota transplantation (FMT) using stool from a donor with low proteolytic activity and containing the bacteria Alistipes putredinis in patients with irritable bowel syndrome (IBS) and high proteolytic activity. Proteolytic activity is the breakdown of proteins into smaller polypeptides or amino acids.

ELIGIBILITY:
Inclusion Criteria:

* IBS defined by Rome IV criteria
* Non IBS-C
* Moderate to severe symptoms defined by IBS-SSS≥175
* Able to safely undergo and consent to colonoscopy

Exclusion Criteria

* Immune deficiency or treatment with immunosuppressive medications
* Severe bowel or medical disease precluding administration of bowel prep
* Severe bowel or medical disease precluding colonoscopy with conscious sedation
* Active cancer
* Pregnant or lactating
* Abdominal surgery (exception of splenectomy, partial hepatectomy, partial/unilateral nephrectomy, laparoscopy, pelvic floor repair, mesh, liposuction, fundoplication, tubal ligation, gastric sleeve, oophorectomy, hernia, appendectomy, cholecystectomy, caesarean section and hysterectomy)
* Severe psychiatric disorder (HADS-A or D>16), or diagnosed alcohol or drug abuse disorder
* New probiotics or treatment with antibiotics, NSAIDs (within 4 wks prior to study entry)
* Use of treatments known to affect colonic motility (with exception of loperamide)
* Diagnosed h/o bleeding disorder
* Organic GI diseases (IBD, celiac disease, microscopic colitis)
* Chronic kidney or liver disease
* Absolute neutrophil count (ANC) <500 IU/ml

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of responders | 12 weeks
  Number of subjects receiving the donor fecal microbiota transplantation identified as a responder defined as a decrease of ≥50 points in Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) from baseline.
  The Irritable Bowel Syndrome Symptom Severity Score scale has a possible range of scores from 0-500. Mild cases are classified as a score of 75-175, moderate cases are classified as a score of 175-300, and severe cases are classified as a score of >300.

SECONDARY OUTCOMES:
Change in level of fecal proteolytic activity | Baseline, 12 weeks
  The level of fecal proteolytic activity will be measured at baseline and again at 12 weeks. The proteolytic activity is measured using a standardized FITC Casein assay that relies on the activity of proteases in the sample to digest casein protein.
Changes in in vivo excretion of 2-24 hr lactulose excretion | Baseline, 12 weeks
  Measured by permeability testing
Number of weekly responders | 12 weeks
  Number of subjects to meet responder criteria of ≥30% decrease in average of worst abdominal pain in past 24 hours plus ≥50% decrease in the number of days per week with at least one stool that has a consistency of Type 6 or 7 (compared with baseline)
Global Adequate Relief Questionnaire | 12 weeks
  Number of subjects to report adequate relief of IBS symptoms, measured by answering yes to question "In the past 7 days have you had adequate relief of your IBS symptoms?"
Alistipes putredinis proportion post-FMT | 12 weeks
  Number of subject to have the bacteria Alistipes putredinis in stool sample after fecal microbiota transplantation (FMT)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials